CLINICAL TRIAL: NCT05899608
Title: A Randomized, Double-blind, Multiregional Phase 3 Study of Ivonescimab Combined With Chemotherapy Versus Pembrolizumab Combined With Chemotherapy for the First-line Treatment of Metastatic Non-small Cell Lung Cancer (HARMONi-3)
Brief Title: Clinical Study of Ivonescimab for First-line Treatment of Metastatic NSCLC Patients
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Summit Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SMT112-3003
Record Dates: First submitted 2023-06-01; First posted 2023-06-12 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A - Ivonescimab and chemotherapy (Experimental): Subject will receive ivonescimab and chemotherapy
  Interventions: Biological: Ivonescimab Injection
- Arm B - Pembrolizumab and chemotherapy (Active Comparator): Subject will receive pembrolizumab and chemotherapy
  Interventions: Biological: Pembrolizumab Injection

INTERVENTIONS:
Biological: Ivonescimab Injection — Subject will receive ivonescimab and chemotherapy as an IV injection
  Arms: Arm A - Ivonescimab and chemotherapy
Biological: Pembrolizumab Injection — Subject will receive pembrolizumab and chemotherapy as an IV injection
  Arms: Arm B - Pembrolizumab and chemotherapy

SUMMARY:
This is a Phase 3 Randomized, double-blind, Multiregional Study of Ivonescimab Combined with Chemotherapy Versus Pembrolizumab Combined with Chemotherapy for the First-line Treatment of Metastatic Non-small Cell Lung Cancer. The primary endpoint is overall survival and progression free survival assessed by investigator. The key secondary endpoints include response and safety.

DETAILED DESCRIPTION:
This study consists of two distinct NSCLC histology cohorts: squamous (N=600) and non-squamous (N=1000), approximately 1600 patients in total. Within each cohort, subjects are randomized in a 1:1 ratio into one of two treatment groups, receiving either ivonescimab or pembrolizumab combined with platinum-doublet chemotherapy. The two histology cohorts will be analyzed independently

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old at the time of enrollment
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1
* Expected life expectancy ≥ 3 months
* Metastatic (Stage IV) NSCLC
* Histologically or cytologically confirmed squamous or non-squamous NSCLC
* Recorded measurement of the Tumor Proportion Score (TPS) or Tumor Cells (TC) for PD-L1 expression, irrespective of the PD-L1 expression, prior to randomization
* At least one measurable noncerebral lesion according to RECIST 1.1
* No prior systemic treatment for metastatic NSCLC

Exclusion Criteria:

* Histologic or cytopathologic evidence of the presence of small cell lung carcinoma
* Known actionable genomic alterations (EGFR, ALK, ROS1, and BRAF V600E) or genes for which first-line approved therapies are available.

  * For non-squamous histology patients, actionable driver mutation testing results are required before randomization.
* Has received any prior therapy for NSCLC in the metastatic setting
* Tumor invasion, encasement of organs (e.g. pericardium, heart, trachea, esophagus, central bronchi), or major blood vessels (e.g aorta, central veins), if poses a significant increased risk of bleeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1600 (Estimated)
Dates: Start 2023-10-26 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | approximately 4 years
  Overall Survival (OS) in the ITT population
Progression Free Survival (PFS) | approximately 3 years
  Progression Free Survival (PFS) assessed by investigator based on RECIST V1.1

SECONDARY OUTCOMES:
Adverse Event (AE) | From the subject signs the ICF to 30 days (AE) and 90 days (SAE related to ivonescimab/pembrolizumab ) after the last dose of study treatment or initiation of other anticancer therapy, whichever occurs first, up to 2 years.
  incidence and severity of adverse events (AEs) and clinically significant abnormal laboratory test results

CONTACTS AND LOCATIONS:
Overall Officials: Indu Lal, Study Director — Summit Therapeutics, Inc.
Locations (244):
- United States (71):
  - Banner University Medical Center, Phoenix, Arizona
  - TMC Healthcare, Tucson, Arizona
  - University of Arkansas, Little Rock, Arkansas
  - LA Cancer Network, Anaheim, California
  - The Oncology Institute of Hope & Innovation, Cerritos, California
  - University of Southern California (USC), Los Angeles, California
  - Cedar Sinai Medical Center, Los Angeles, California
  - Valkyrie Clinical Trials, Los Angeles, California
  - Sutter Institute for Medical Research, Sacramento, California
  - UC Davis Medical Center, Sacramento, California
  - University of California Los Angeles (UCLA), Santa Monica, California
  - Providence Medical Foundation, Santa Rosa, California
  - Kaiser Permanente, Vallejo, California
  - Rocky Mountain Cancer, Lone Tree, Colorado
  - Banner MD Anderson Cancer Center at North Colorado Medical Center, Loveland, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Florida Cancer Specialists & Research Institute (FCS)-East, Fort Myers, Florida
  - BioResearch Partner- Hialeah Hospital, Hialeah, Florida
  - Mayo Clinic, Jacksonville, Florida
  - Cancer Specialists of North Florida, Jacksonville, Florida
  - Ocala Oncology, Ocala, Florida
  - Cancer Care of Brevard, Palm Bay, Florida
  - Memorial Cancer Institute, Pembroke Pines, Florida
  - Ascension Sacred Heart Health System, Pensacola, Florida
  - Exigent Network, Petersburg, Florida
  - BRCR Medical Center Inc, Plantation, Florida
  - Florida Cancer Specialists & Research Institute (FCS) - North, St. Petersburg, Florida
  - BRCR Medical Center Inc., Tamarac, Florida
  - Florida Cancer Specialists & Research Institute (FCS)-South, West Palm Beach, Florida
  - Illinois Cancer Care, Peoria, Illinois
  - University of Kansas Cancer Center, Westwood, Kansas
  - Baptist Health, Lexington, Kentucky
  - Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Ascension Saint Agnes Hospital, Baltimore, Maryland
  - Lahey Hospital, Burlington, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Trinity Health, Ann Arbor, Michigan
  - Karmanos Cancer Insitute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Park Nicollet Institute, Saint Paul, Minnesota
  - American Oncology Partners, PA, Kansas City, Missouri
  - Washington University St.Louis, St Louis, Missouri
  - St. Vincent Cancer Center, Billings, Montana
  - University of Nebraska Medical Center (UNMC), Omaha, Nebraska
  - Mount Sinai, New York, New York
  - Memorial Sloan Kettering, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Levine Center, Charlotte, North Carolina
  - Oncology Hematology Care (OHC), Inc, Cincinnati, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Willamette Valley Cancer Institute and Research Center (WVCI), Eugene, Oregon
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Prisma Health-Upstate, Greenville, South Carolina
  - West Cancer Center, Memphis, Tennessee
  - SCRI-Nashville, Nashville, Tennessee
  - Texas Oncology- Austin, Austin, Texas
  - Texas Oncology-Dallas, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Texas Oncology-San Antonio, San Antonio, Texas
  - Texas Oncology-Tyler, Tyler, Texas
  - University of Texas at Tyler, Tyler, Texas
  - Virginia Oncology Associates, Norfolk, Virginia
  - Virginia Cancer, Reston, Virginia
  - Swedish Cancer Institute, Seattle, Washington
  - Cancer Care NW Centers, Spokane, Washington
  - Carbone Cancer Center, Madison, Wisconsin
- Belgium (2):
  - CHU UC Louvain Namur, Louvain-la-Neuve
  - az Glorieux, Ronse
- Canada (3):
  - London Regional (LRCP), London, Ontario
  - Ottawa Cancer Center, Ottawa, Ontario
  - Saskatchewan Cancer, Regina, Saskatchewan
- China (45):
  - Fu Yang People's Hospital, Yangzhou, Anhui
  - Beijing Chest Hospital, Tongzhou, Beijing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Gansu Provincial Cancer Hospital, Lanzhou, Gansu
  - Fujian Cancer Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Hainan General Hospital, Haikou, Hainan
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan University of Science and Technology Affiliated Anyang Cancer Hospital, Anyang, Henan
  - Nanyang Central Hospital, Nanyang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Henan University of Science and Technology Affiliated Anyang Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Yangtze University, Jingzhou, Hubei
  - Xiangyang Central Hospital, Xiangyang, Hubei
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - Hunan Cancer Hospital Thoracic Medicine 1, Changsha, Hunan
  - The First Affiliated Hospital Of University Of South China, Hengyang, Hunan
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - First Affiliated Hospital of Gannan Medical University, Ganzhou, Jiangxi
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Jiangxi Cancer Hospital, Nanchang, Jiangxi
  - Shengjing Hospital Of China Medical University, Shenyang, Liaoning
  - The Second Affiliated Hospital of AFMU, Xi'an, Shaanxi
  - The first affiliated Hospital of xi'an jiao tong university, Xi'an, Shaanxi
  - Shandong Cancer Hospital, Jinan, Shandong
  - Linyi People's Hospital, Linyi, Shandong
  - Qingdao Central Hospital, Qingdao, Shandong
  - Fudan University Shanghai Cancer Center, Xuhui, Shanghai Municipality
  - Shanghai Chest Hospital, Xuhui, Shanghai Municipality
  - Shanghai Pulmonary Hospital, Yangpu, Shanghai Municipality
  - Shanxi Provincial Cancer Hospital, Taiyuan, Shanxi
  - Mianyang Central Hospital, Mianyang, Sichuan
  - Cancer Hospital Affiliated to Xinjiang Medical University, Ürümqi, Xinjiang
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - The First Affiliated Hospital,Zhejiang University, Hanzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hanzhou, Zhejiang
  - Jinhua Municipal Central Hospital, Jinhua, Zhejiang
  - Ningbo Medical Center Lihuili Hospital, Ningbo, Zhejiang
  - TaiZhou Hospital Of Zhejiang Province, Taizhou, Zhejiang
  - Cancer Hospital Chinese Academy of Medical Science, Beijing
  - Peking University People's Hospital, Beijing
  - The Fifth Medical Center of the General Hospital of the Chinese People's Liberation Army, Beijing
  - Hunan Cancer Hospital Thoracic Medicine 2, Changsha
  - Guangxi Medical University Cancer Hospital, Guangxi
- France (15):
  - Centre Hospitalier Regional Universitaire (CHRU) Brest, Brest
  - Centre Hospitalier Universitaire (CHU) de Caen, Caen
  - Unicancer - Centre François Baclesse (CFB), Caen
  - Centre Hospitalier Intercommunal de Creteil (CHIC, Créteil
  - Centre de Cancérologie de la Sarthe, Le Mans
  - Hopital Nord, Marseille
  - Centre Hospitalier Universitaire de Montpellier (CHU Montpellier), Montpellier
  - Institut Curie, Paris
  - Centre Hospitalier Lyon-Sud, Pierre-Bénite
  - Centre Hospitalier (Intercommunal) De Cornouaille Quimper, Quimper
  - Centre Hospitalier Universitaire (CHU) de Rennes, Rennes
  - Institut de Cancérologie de l'Ouest, Saint-Herblain
  - Institut de cancérologie Strasbourg Europe (ICANS), Strasbourg
  - Centre Hospitalier Regional et Universitaire de Tours, Tours
  - Gustave Roussy Oncologie Médical, Villejuif
- Germany (9):
  - Klinikum Esslingen GmbH, Esslingen am Neckar
  - Krankenhaus Nordwest GmbH, Frankfurt
  - Asklepios Klinik Gauting GmbH, Gauting
  - Universitaetsklinikum Giessen und Marburg, Giesen
  - Universitaetsklinikum Heidelberg (UKHD), Heidelberg
  - Universitaetsklinikum Jena, Jena
  - Klinikverbund Allgaeu - Klinikum Kempte, Kempten
  - Universitätsklinikum Schleswig-Holstein, Lübeck
  - München Klinik gGmbH, Munich
- Greece (9):
  - Henry Dunant Hospital Center, Athens
  - General Hospital of Athens, Athens
  - General Hospital of Athens Alexandra, Athens
  - Metropolitan General Hospital, Athens
  - Interbalkan Medical Center of Thessaloniki, Athens
  - Olympion Hospital, Pátrai
  - University General Hospital of Patras, Pátrai
  - Galenos General Clinic, Thessaloniki
  - "George Papanikolaou" General Hospital of Thessaloniki, Thessaloniki
- Ireland (3):
  - St. James's Hospital (SJH), Dublin
  - Beaumont Hospital, Dublin
  - Galway Univeristy Hospitals, Galway
- Italy (15):
  - Azienda Ospedaliero Universitaria delle Marche, Ancona
  - Centro di Riferimento Oncologico di Aviano, Aviano
  - Azienda Ospedaliera "Istituti Ospitalieri" di Cremona, Cremona
  - Istituto Europeo di Oncologia (IEO), Genova
  - Ospedale San Luca, Lucca
  - Fondazione IRCCS - Istituto Nazionale dei Tumori - Milano, Milan
  - Istituto Europeo di Oncologia (IEO), Milan
  - Fondazione IRCCS San Gerardo dei Tintori, Monza
  - Universita degli Studi della Campania "Luigi Vanvitelli", Naples
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Azienda Sanitaria Territoriale Pesaro Urbino (AST PU), Pesaro
  - Ospedale P. Pederzoli, Peschiera del Garda
  - Istituti Fisioterapici Ospitalieri (IFO), Roma
  - Azienda Ospedaliera Universitaria Senese - Istituto Toscano Tumori, Siena
  - Ospedale G.B. Rossi Borgo Roma, Verona
- Japan (18):
  - Fujita Health University Hospital, Aichi
  - National Hospital Organization Kyusyu Medical Center, Fukuoka
  - Hirosaki University Hospital, Hirosaki
  - Hiroshima University Hospital, Hiroshima
  - National Hospital Organization - Hokkaido Cancer Center, Hokkaido
  - Hakodate Goryoukaku Hospital, Hokkaido
  - Nara Medical University Hospital, Kashihara
  - Shinshu University Hospital, Matsumoto
  - Sendai Kousei Hospital, Miyagi
  - Okayama University Hospital, Okayama
  - Osaka Medical and Pharmaceutical University Hospital (OMPU Hp), Osaka
  - Kansai Medical University Hospital, Osaka
  - Shizuoka Cancer Center (SCC), Shizuoka
  - National Cancer Center Hospital (NCCH), Tokyo
  - The Cancer institute Hospital, Tokyo
  - National Hospital Organization Yamaguchi Ube Medical Center, Yamaguchi
  - Kanagawa Cancer Center, Yokohama
  - Tottori University Hospital, Yonago
- Mexico (12):
  - Panamerican Clinical Research S.A de C.V., Guadalajara
  - Actualidad Basada en Investigación del Cáncer, Guadalajara
  - Renati Innovation S.A.P.I. DE C.V., Guadalajara
  - Centro de Atención Oncológica Viva, La Paz
  - Health Pharma Professional Research S.A. de C.V., Mexico City
  - Centro de Investigación Clínica GRAMEL, Mexico City
  - Arke SMO S.A DE C.V, Mexico City
  - Centro de Atención Oncológica Viva, Mexico City
  - Althian Clinical Research, Monterrey
  - CRI Centro Regiomontano de Investigación S.C., Monterrey
  - Hospital Universitario "Dr. José Eleuterio González", Monterrey
  - I Can Oncology Center, Monterrey
- Poland (5):
  - Centrum Onkologii im. prof. F. Lukaszczyka w Bydgoszczy, Bydgoszcz
  - Instytut Msf Sp. z o.o., Lodz
  - Med Polonia Sp. z o.o. NSZOZ, Poznan
  - Szpital Specjalistyczny w Prabutach, Prabuty
  - Wojskowy Instytut Medczny, Warsaw
- Serbia (7):
  - Acibadem Bel Medic General Hospital, Belgrade
  - Klinicki Centar Srbije, Belgrade
  - Vojnomedicinska Akademija (VMA), Belgrade
  - Klinicko Bolnicki Centar (KBC) Bezanijska Kosa, Belgrade
  - Institut Za Plucne Bolesti Vojvodine Klinika za pulmolosku onkologiju, Kamenica
  - Univerzitetski Klinicki Centar Kragujevac, Kragujevac
  - University Clinical Center Niš, Niš
- Spain (19):
  - Hospital Universitario de Badajoz, Badajoz
  - Hospital Universitari Germans Trias i Pujol, Badalona
  - Instituto Oncologico Baselga (IOB), Barcelona
  - Hospital de la Santa Creu i de Sant Pau, Barcelona
  - Hospital Universitari Dexeus, Barcelona
  - Vall d'Hebron University, Barcelona
  - Mi Tres Torres, Barcelona
  - Institut d'Investigacio Biomedica de Girona Dr. Josep Trueta, Girona
  - Hospital Universitario de Jaén, Jaén
  - Universidad de Las Palmas de Gran Canaria, Las Palmas de Gran Canaria
  - Hospital Universitario Lucus Augusti (HULA), Lugo
  - Universidad Autonoma de Madrid (UAM), Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Regional Universitario de Málaga, Málaga
  - Clinica Universidad de Navarra (CUN) - Pamplona, Pamplona
  - H Universitario Virgen Del Rocio, Seville
  - Hospital Clinico Universitario de Valencia (CHUV), Valencia
  - Hospital La Fe Bulevar Sur, Valencia
  - Hospital Alvaro Cunqueiro (HAC), Vigo
- Sweden (2):
  - Karolinska University Hospital, Stockholm
  - Region Gävleborg Gävle Sjukhus Gävle Sjukhus, Uppsala
- Turkey (Türkiye) (6):
  - Memorial Ankara Hospital, Ankara
  - Dicle University, Diyarbakır
  - Memorial Saglik Grubu Bahçelievler Hospital, Istanbul
  - Istinye University Bahceshir Liv Hospital, Istanbul
  - Kocaeli University Hospital, İzmit
  - Necmettin Erbakan University Meram Medical Faculty Hospital, Konya
- United Kingdom (3):
  - Leeds Teaching Hospitals NHS, Leeds
  - St. Bartholomew's hospital, London
  - The Christie NHS Foundation Trust, Manchester